CLINICAL TRIAL: NCT02685267
Title: A Phase II Randomized Prospective Trial of Docetaxel/Prednisone Versus Docetaxel/Prednisone and Enzalutamide in Castration-Resistant Prostate Cancer (CRPC) Patients Progressing on Enzalutamide
Brief Title: Docetaxel/Prednisone Versus Docetaxel/Prednisone and Enzalutamide in Castration-Resistant Prostate Cancer
Acronym: Doce/Enza
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Prostate Cancer Clinical Trials Consortium (Other)
Collaborators: University of Chicago (Other); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: c13-126
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; enzalutamide; Prednisone

ARMS (2):
- Docetaxel/Prednisone (Active Comparator): Docetaxel 75 mg/m2 day 1 (every 21-days) plus prednisone 5 mg po bid throughout
  Interventions: Drug: Docetaxel; Drug: Prednisone
- Docetaxel/Prednisone + Enzalutamide (Active Comparator): Docetaxel 75 mg/m2 day 1 (every 21-days) plus prednisone 5 mg po bid throughout plus Enzalutamide 160 mg daily throughout. Subjects will continue enzalutamide until PD after 10 cycles of docetaxel.
  Interventions: Drug: Docetaxel; Drug: Enzalutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel
Drug: Enzalutamide
  Arms: Docetaxel/Prednisone + Enzalutamide
Drug: Prednisone

SUMMARY:
This is a prospective randomized phase II clinical trial where patients who are receiving enzalutamide in the pre-chemotherapy space are randomized upon objective progression (radiographic and/or clinical per PCWG2 criteria) to docetaxel/prednisone alone or the same combination plus enzalutamide.

The primary aim is to evaluate whether continuing enzalutamide in combination with docetaxel in patients who failed or progressed while on enzalutamide would increase progression-free survival (PFS) by 4 months. The secondary end points are PSA responses, percent of patients alive at 1 and 2 years, decline in circulating tumor cells (CTCs), and quality of life (QOL) using validated scales.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.

NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.

* Males 18 years of age and above
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Having documented disease progression on enzalutamide defined by 1 or more of the following criteria:
* PSA progression according to PCWG2 criteria with 3 consecutive rising PSA measurements, all collected at least 1 week apart
* Radiographic progression in soft tissue or bone by modified RECIST 1.1 for subjects with measurable disease; or
* Bone disease progression defined by 2 or more new lesions on 2 consecutive bone scans in the absence of falling PSA
* Patients who have not had a bilateral orchiectomy must have a plan to maintain effective GnRG-analogue therapy for the duration of the trial
* Serum testosterone level < 50 ng/dL at Screening visit
* ECOG PS: 0-1
* Throughout the study, male patients and their female partners of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration. Two acceptable methods of birth control thus include the following:
* Condom (barrier method of contraception even if having sex with a pregnant woman)
* One of the following is required:

  * Established use of oral, injected, or implanted hormonal method of contraception by the female partner
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner
  * Additional barrier method: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female partner
  * Tubal litigation in the female partner
  * Vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy) for >6 months
* Patients must have adequate organ and marrow function as defined below
* Leukocytes >3,000/mm3
* absolute neutrophil count >1,500/mm3
* platelets >100,000/mm3
* total bilirubin within normal institutional limits (or <2X the upper limit of normal in those with Gilbert's disease)
* AST(SGOT)/ALT(SGPT) <1.5 X institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance* >45 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Estimated life expectancy of > 6 months
* Able to swallow the study drug as prescribed and comply with study requirements

Exclusion Criteria:

* Prior treatment with docetaxel-based chemotherapy
* Prior treatment with abiraterone acetate
* Prior treatment with cabazitaxel
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment
* Ongoing investigational treatment
* Medical conditions such as uncontrolled hypertension, uncontrolled diabetes mellitus, cardiac disease that would, in the opinion of the investigator, make this protocol unreasonably hazardous
* Major surgery within 4 weeks of enrollment
* Use of an investigational therapeutic agent with 4 weeks of enrollment
* History of seizure or any condition that may predispose to seizure.
* History of loss of consciousness or transient ischemic attack within 12 months of enrollment
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease) within last 3 months
* Grade > 2 treatment-related toxicity from prior therapy
* History of hypersensitivity to polysorbate 80
* Any known allergy to the compounds under investigation
* Any other condition which, in the opinion of the Investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSytem - Kellogg Cancer Center, Evanston, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Univesity of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel/Prednisone: Docetaxel 75 mg/m2 day 1 (every 21-days) plus prednisone 5 mg po bid throughout
  Docetaxel
  Prednisone
- Docetaxel/Prednisone + Enzalutamide: Docetaxel 75 mg/m2 day 1 (every 21-days) plus prednisone 5 mg po bid throughout plus Enzalutamide 160 mg daily throughout. Subjects will continue enzalutamide until PD after 10 cycles of docetaxel.
  Docetaxel
  Enzalutamide
  Prednisone
Period: Overall Study
Arm/Group | Docetaxel/Prednisone | Docetaxel/Prednisone + Enzalutamide
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel/Prednisone | Docetaxel/Prednisone + Enzalutamide | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 68.2 [55 to 84] | 67.25 [58 to 79] | 67.78 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (Radiographic or Per PCWG2 Criteria)
Description: The primary endpoint of the study is progression-free survival (PFS), defined as the time from randomization to disease progression. Progression will be evaluated using a combination of RECIST and Prostate Cancer Working Group 2 guidelines.
Time Frame: 1 year
Population: As the study was terminated after only 9 patients enrolled, 5 to the standard of care docetaxel/prednisone arm and 4 to experimental docetaxel/prednisone/enzalutamide arm, the study was not evaluable for any efficacy endpoints.
  Sufficient data for the primary endpoint were not collected to provide outcome measures data tables below.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel/Prednisone | Docetaxel/Prednisone + Enzalutamide
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0
Statistical Analysis 1: Comparison: Docetaxel/Prednisone; The study was terminated after only 9 patients enrolled, 5 to the standard of care docetaxel/prednisone arm and 4 to experimental docetaxel/prednisone/enzalutamide arm; Test type: Other — The study was terminated after only 9 patients enrolled, 5 to the standard of care docetaxel/prednisone arm and 4 to experimental docetaxel/prednisone/enzalutamide arm; p = 0.6761, Chi-squared; log-rank test = 0.6761

2. Secondary Outcome: PSA Response in the Standard Treatment Arm and Experimental Treatment Arm
Description: PSA response measured according to Prostate Cancer Working Group 2 (PCWG2).
  The study was terminated after only 9 patients enrolled, 5 to the standard of care docetaxel/prednisone arm and 4 to experimental docetaxel/prednisone/enzalutamide arm.
Time Frame: Baseline, Day 84 (C4D1), Day 147 (C7D1), Day 210 (C10D1), Day 231, and every 21 days through study completion (an average of 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel/Prednisone | Docetaxel/Prednisone + Enzalutamide
Number analyzed (Participants) | 5 | 4
Participants | 2 | 3

3. Secondary Outcome: Overall Survival
Time Frame: At both 1 year and 2 years from treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel/Prednisone | Docetaxel/Prednisone + Enzalutamide
Number analyzed (Participants) | 5 | 4
Participants | 2 | 4

4. Other Pre Specified Outcome: Quality of Life (QOL)
Time Frame: Baseline, Day 84 (C4D1), Day 147 (C7D1), Day 210 (C10D1), Day 231 and every 21 days through study completion (an average of 1 year)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Circulating Tumor Cells (CTCs)
Time Frame: Baseline, Day 84 (C4D1), Day 147 (C7D1), Day 210 (C10D1), and every 63 days through study completion (an average of 1 year)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Analysis of Androgen Receptor Splice Variant
Time Frame: as for outcome 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From treatment administration through 30 days after date of last dose
Arm/Group | Docetaxel/Prednisone | Docetaxel/Prednisone + Enzalutamide
All-Cause Mortality (participants affected / at risk) | 3/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel/Prednisone (N=5) | Docetaxel/Prednisone + Enzalutamide (N=4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel/Prednisone (N=5) | Docetaxel/Prednisone + Enzalutamide (N=4)
Fatigue (General disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Edema limbs (Blood and lymphatic system disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Blood and lymphatic system disorders) | 1 | 0
Watering eyes (Eye disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Left great toe pain (Skin and subcutaneous tissue disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Bell's Palsy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye infection (Eye disorders) | 0 | 1
Lacrimation (Eye disorders) | 0 | 1
Nail pain (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT02685267/Prot_SAP_000.pdf